CLINICAL TRIAL: NCT00399659
Title: A 52-week Extension to Study CHTF919N2201 to Evaluate the Safety and Efficacy of Tegaserod (6 mg b.i.d. and 12 mg o.d.) Given Orally for the Treatment of Opioid-induced Constipation (OIC) in Patients With Chronic Non-cancer Pain
Brief Title: Safety and Efficacy of Tegaserod in Opioid-induced Constipation in Patients With Non-cancer Pain.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early as a result of regulatory action suspending tegaserod use in 2007
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919N2201E1
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid, constipation, tegaserod
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study will evaluate the safety and efficacy of Tegaserod in opioid-induced constipation (OIC) in patients with non-cancer pain.

Patients who enter this study PRIOR to the core study (CHTF919N2201) interim analysis (IA) receive the treatment as follows:

Patients on tegaserod 6 mg twice daily (b.i.d.) or 12 mg once daily (o.d.) in the core study will remain on the same dose in the extension (double-blind).

Patients on placebo during the core study will receive tegaserod 12 mg o.d. (open-label)

Patients who enter this study AFTER the core study interim analysis will receive the selected tegaserod dose regimen (open-label) determined by the core study IA.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed the 12 week double blind treatment of study CHTF919N2201

Exclusion Criteria:

* Planned discontinuation of opioids during the study.
* Development of any of the medical conditions listed as exclusion criteria for the CHTF919N2201 study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Long term safety of tegaserod

SECONDARY OUTCOMES:
Change from baseline assessment of OIC symptoms, at week 24 and 52
Change from baseline assessment of opioid-induced mid/upper GI symptoms, at week 24 and 52
Patients' weekly assessment of intensity of pain for which opioids were prescribed, at week 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corp., Study Chair — NPC
Locations (52):
- United States (52):
  - Investigative Site, Mobile, Alabama
  - Investigative Site, Phoenix, Arizona
  - Investigative Site, Tucson, Arizona
  - Investigative Site, North Little Rock, Arkansas
  - Investigative Site, Buena Park, California
  - Investigative Site, Downey, California
  - Investigative Site, Encinitas, California
  - Investigative Site, Fountain Valley, California
  - Investigative Site, La Jolla, California
  - Investigative Site, Los Angeles, California
  - Investigative Site, Mission Viejo, California
  - Investigative Site, Monroe, California
  - Investigative Site, San Diego, California
  - Investigative Site, San Francisco, California
  - Investigative Site, Torrance, California
  - Investigative Site, Northglenn, Colorado
  - Investigative Site, Bristol, Connecticut
  - Investigative Site, DeLande, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Largo, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, New Smyrna Beach, Florida
  - Investigative Site, Sarasota, Florida
  - Investigative Site, Springhill, Florida
  - Investigative Site, Tampa, Florida
  - Investigative Site, Belleville, Illinois
  - Investigative Site, Chicago, Illinois
  - Investigative Site, Avon, Indiana
  - Investigative Site, Evansville, Indiana
  - Investigative Site, Indianapolis, Indiana
  - Investigative Site, Overland Park, Kansas
  - Investigative Site, Prairie Village, Kansas
  - Investigative Site, Topeka, Kansas
  - Investigative Site, Shreveport, Louisiana
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Wellesley Hills, Massachusetts
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Pahrump, Nevada
  - Investigative Site, New York, New York
  - Investigative Site, North Massapequa, New York
  - Investigative Site, Charlotte, North Carolina
  - Investigative Site, Greensboro, North Carolina
  - Investigative Site, Winston-Salem, North Carolina
  - Investigative Site, Oklahoma City, Oklahoma
  - Investigative Site, Levittown, Pennsylvania
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Beaumont, Texas
  - Investigative Site, Corsicana, Texas
  - Investigative Site, Houston, Texas
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Charlottesville, Virginia
  - Investigative Site, Seattle, Washington